CLINICAL TRIAL: NCT05383027
Title: Examining the Feasibility of Implementation, Patterns of Association, and Outcomes in HRV Biofeedback (HRVB) Intervention and Music Listening Control (MLC) on Alzheimer's Disease (AD) Family Caregivers (FCGs) Public Title: Caring Relationship Expression Study(CARES)
Brief Title: Examining the Feasibility of Implementation, Patterns of Association, and Outcomes in HRV Biofeedback (HRVB) Intervention and Music Listening Control (MLC) on Alzheimer's Disease (AD) Family Caregivers (FCGs) Public Title: Caring Relationship Expression Study
Acronym: CARES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 000141913
Record Dates: First submitted 2022-05-17; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer's Disease and Related Dementias Family Caregivers
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Listening Control(MLC) (Active Comparator)
  Interventions: Behavioral: Music Listening Control (MLC)
- Heart Focused Breathing (Experimental)
  Interventions: Behavioral: Heart Focused Breathing

INTERVENTIONS:
Behavioral: Music Listening Control (MLC) — MLC participants will engage in assigned music listening in the presence of their loved one with ADRD via a selected online platform (pandora or Spotify) for 10 minutes a day 5-7 days a week.
  Arms: Music Listening Control(MLC)
Behavioral: Heart Focused Breathing — Heart-focused breathing participants will engage in heart-focused breathing using the inner balance device (shipped to their home), they will be asked to do this in the presence of their loved one with ADRD for 10 minutes a day 5-7 days per week.
  Arms: Heart Focused Breathing

SUMMARY:
In a remotely delivered nationwide pilot study, we will be examining a novel 8-week heart rate variability biofeedback (HRVB) intervention vs music listening control (MLC) for 30 family caregivers 18 years and older (FCGs) of Alzheimer's disease (AD) (and related dementias: ADRD) patients to examine feasibility (acceptability/adherence, satisfaction) and direction of change in caregiver burden, stress, resilience, anxiety, self-compassion, and relationship quality.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above
* primary, unpaid family caregiver for ADRD patient for 6 months or more
* owns and operates a smartphone with a data plan
* greater than of equal to 4 on caregiver burden scale

Exclusion Criteria:

* regular mind-body practice
* under 18 years old
* pacemaker
* conditions or medications that interfere with heart rate variability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale-10 | 13 weeks
  Measure of stress
Zarit Burden Interview | 13 weeks
  Measures participant burden
Brief Resilience Scale | 13 weeks
  Measures participant resillience

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided